CLINICAL TRIAL: NCT04864977
Title: Novel Approach for Basal Insulin Titration: A Proof-of-Concept Study
Brief Title: A Study of A Novel Approach to Titrate Basal Insulin (LY2963016) in Participants With Type 2 Diabetes
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Study was stopped prior to study start date due to business decision.
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18095; I4L-MC-YCAA (Other: Eli Lilly and Company)
Record Dates: First submitted 2021-04-27; First posted 2021-04-29 (Actual); Last update posted 2021-08-24 (Actual); Status verified 2021-08

CONDITIONS: Type 2 Diabetes; Type 2 Diabetes Treated With Insulin
Keywords: T2D
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — LY2963016 insulin glargine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- LY2963016 (Experimental): Participants with type 2 diabetes will be started on insulin glargine and dose will be titrated. Insulin glargine will be delivered via insulin pen each evening subcutaneously (SC). They will also check fasting blood glucose values on a study meter and prior to treating hypoglycemia. Participants will be asked to report the time and dose of their last administration.
  Interventions: Drug: Basal Insulin

INTERVENTIONS:
Drug: Basal Insulin — Participants administered basal insulin
  Other Names: LY2963016

SUMMARY:
The main purpose of this study is to evaluate a novel approach for insulin glargine (LY2963016) titration for insulin-naïve adults with type 2 diabetes (T2D)

The study will last about 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Adults with type 2 diabetes as diagnosed by endocrinologist
* No insulin over past 3 months
* Inadequate glycemic control with A1c ≥8.0% at or within 1 month prior to screening visit
* No history of diabetic ketoacidosis (DKA) or severe hypoglycemia leading to mental status change in the past 6 months
* Willingness and ability to follow the protocol including willingness to commence basal insulin, wear CGM, and communicate with healthcare provider.

Exclusion Criteria:

* Contraindication to use of insulin glargine (e.g., allergy)
* Impaired recognition of hypoglycemia by the participant (as judged by the investigator)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-08-16 (Estimated); Primary Completion 2022-06-06 (Estimated); Study Completion 2022-06-06 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants with Type 2 Diabetes Who Achieve Nadir Glucose in Range 70-125 milligram/deciliter (mg/dL) | Week 12
  Percentage of participants with type 2 diabetes who achieve nadir glucose in range (70-125 mg/dl) over 15 consecutive minutes for ≥70% of days (typically 10 days) (last 14 days of active treatment)

SECONDARY OUTCOMES:
Percentage of Participants with Hemoglobin A1c (HbA1c) at target (<7.0%) | Week 12
Percentage of Participants with time in range (TIR) 70-180 mg/dl ≥70% | Week 12
Percentage of Participants who successfully use Continuous Glucose Monitoring (CGM) | Week 12

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, CSR
Time Frame: data are available 6 months after the primary publication and approval of the indication studied in the US and European Union (EU), whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: http://vivli.org/

REFERENCES:
- See also: A Study of A Novel Approach to Titrate Basal Insulin (LY2963016) in Participants With Type 2 Diabetes — https://trials.lillytrialguide.com/en-US/trial/4QTvp0wrJ1GiK4youuzfmY